CLINICAL TRIAL: NCT04518709
Title: The Effect of Posterior Annulus Elevation Technique in Reducing Residual Regurgitation During Mitral Valve Repair in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Cardiovascular Center Harapan Kita Hospital Indonesia (Other)
Responsible Party: Principal Investigator, Budi Rahmat, Chief of Pediatric & Congenital Heart Surgery Division, National Cardiovascular Center Harapan Kita Hospital Indonesia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NationalCCHK
Record Dates: First submitted 2020-08-02; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Mitral Valve Insufficiency
Keywords: Posterior Annulus Elevation Technique; Pediatric Mitral Valve Insufficiency
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Posterior Annulus Elevation Technique Group (Experimental): In patients who were determined in the treatment group, after the conventional procedure for mitral valve repair was completed, a posterior mitral valve elevation technique will be performed.
  Interventions: Procedure: Posterior Mitral Annulus Elevation Technique
- Without Posterior Annulus Elevation Technique Group (Placebo Comparator): No additional procedure will be done after conventional mitral valve repair
  Interventions: Procedure: Conventional Mitral Valve Repair

INTERVENTIONS:
Procedure: Posterior Mitral Annulus Elevation Technique — Posterior mitral annulus elevation technique is performed using a large pledget and non-absorbable braided suture starting from the subvalvular section of the posterior mitral valve sutured to the ring annuloplasty (if in the process of repairing the mitral valve, ring implantation is performed; if without the use of ring annuloplasty, the suture is placed in the left atrial wall / supravalvular of PML), so that the posterior annulus is slightly attracted upward toward the cranial and the PML moves toward the center.
  Arms: Posterior Annulus Elevation Technique Group
Procedure: Conventional Mitral Valve Repair — Conventional mitral valve repair in the pediatric patient using annuloplasty, leaflet resection and plication, sliding-plasty of chordae technique
  Arms: Without Posterior Annulus Elevation Technique Group

SUMMARY:
The main problem in mitral valve repair surgery in children is the high number of postoperative residual lesions (49% of the total cases). Residual lesions after mitral valve repair are associated with morbidity and complications in the form of hemolysis and could affect the postoperative reverse remodeling process. Surgery techniques for mitral valve repair in children have fewer choices than adult patients because of the smaller and thinner valve structure. Besides, the weakness of the mitral valve repair technique that often occurs in large left ventricles with severe mitral regurgitation, after repairing with ring annuloplasty, there is usually a mild residual regurgitation due to posterior mitral leaflet that tends to become restrictive due to being attracted by the left ventricular wall that remains big. No technique has been found to overcome the problem of mitral regurgitation residuals that occur postoperatively. Therefore, by analyzing postoperative mitral valve structural abnormalities with conventional techniques, an additional posterior mitral valve elevation technique was designed to increase the area of coaptation between two leaves of the mitral valve so that the incidence of postoperative regurgitation lesions can be reduced.

DETAILED DESCRIPTION:
The main problem in mitral valve repair surgery in children is the high number of postoperative residual lesions (49% of the total cases). Residual lesions after mitral valve repair are associated with morbidity and complications in the form of hemolysis and could affect the postoperative reverse remodeling process. Surgery techniques for mitral valve repair in children have fewer choices than adult patients because of the smaller and thinner valve structure. Besides, the weakness of the mitral valve repair technique that often occurs in large left ventricles with severe mitral regurgitation, after repairing with ring annuloplasty, there is usually a mild residual regurgitation due to posterior mitral leaflet that tends to become restrictive due to being attracted by the left ventricular wall that remains big. No technique has been found to overcome the problem of mitral regurgitation residuals that occur postoperatively.

Therefore, by analyzing postoperative mitral valve structural abnormalities with conventional techniques, an additional posterior mitral valve elevation technique was designed. The posterior annulus elevation technique is a technique that is carried by lifting the posterior mitral annulus towards the cranial so that the posterior mitral leaflet can meet perfectly with the anterior mitral leaflet indicated by a larger coaptation area. This technique can be applied after repair with conventional techniques done optimally to reduce the possibility of postoperative residual lesions.

The hypothesis in this study is that pediatric patients with mitral regurgitation who undergo mitral valve repair surgery with posterior annulus elevation techniques can reduce residual mitral regurgitation, improve clinical and metabolic outcomes of postoperative heart failure, and reduce the risk of postoperative hemolysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with mitral regurgitation heart disease.
2. Patients with an age range of 1 day - 18 years
3. Patients with mitral regurgitation heart disease with atrial septal defects
4. Mitral valve repair surgery performed by single surgeon (Budi Rahmat, MD)

Exclusion Criteria:

1. Patients refuse to participate in the study.
2. Having additional cardiac abnormalities other than atrial septal defects that change the surgery plan.
3. Reoperation mitral valve surgery.
4. History of abnormalities in the central nervous system / preoperative stroke.
5. Patients with severe pulmonary hypertension
6. Patients with small left ventricles (LV smallish)
7. History of pulmonary resuscitation (CPR) before surgery.

Dropout Criteria

1. The patient fails to complete the entire examination procedure.
2. Mitral regurgitation patients who are decided to do mitral valve replacement intra-operatively.
3. Using extracorporeal life support (ECMO) device after surgery.
4. History of intra-operative CPR.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Estimated)
Dates: Start 2020-08-17 (Estimated); Primary Completion 2022-08-17 (Estimated); Study Completion 2022-08-17 (Estimated)

PRIMARY OUTCOMES:
Residual mitral valve regurgitation | 5 days after surgery
  Residual mitral valve regurgitation is measured using transesophageal echocardiography and transthoracic echocardiography
Mitral valve coaptation area | Intraoperative
  Mitral valve coaptation area is measured using transesophageal echocardiography and transthoracic echocardiography
Change of Haptoglobin at 3 months after surgery | Preoperative (baseline), 5 days, 2 weeks and 3 months after surgery
  Serum haptoglobin level that indicated the presence of intravascular hemolysis is measured after the surgery
Change of Lactate dehydrogenase at 3 months after surgery | Preoperative (baseline), 5 days, 2 weeks and 3 months after surgery
  Lactate dehydrogenase level that indicated the presence of intravascular hemolysis is measured after the surgery
Change of NT-proBNP at 3 months after surgery | Preoperative (baseline), 5 days, 2 weeks and 3 months after surgery
  NTproBNP is a marker of acute heart failure and indicates the process of heart remodeling.